CLINICAL TRIAL: NCT00212732
Title: Controlled Study of ONO-8025 (KRP-197) in Patients With Overactive Bladder in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-8025-08
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Overactive Bladder
Keywords: ONO-8025, KRP-197, overactive bladder, antimuscarinic
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — imidafenacin

INTERVENTIONS:
Drug: ONO-8025 (KRP-197)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ONO-8025 (KRP-197) in patients with overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 20 years old or over with overactive bladder
2. Total number of urinary incontinence episodes per week is 5 or over
3. Mean number of micturition per day is 8 or over
4. Mean number of urinary urgency episodes per day is 1 or over
5. Other inclusion criteria as specified in the study protocol

Exclusion Criteria:

1. Patients with genuine stress incontinence
2. Patients suffering from complications such as bladder tumor, bladder stone and urinary tract infection
3. Patients who have undergone surgical operation of urinary and/or genital organs within 6 months prior to the study
4. Patients suffering from complications for which anticholinergics are contraindicated
5. Other exlcusion criteria as specified in the study protocol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750
Dates: Start 2003-10; Primary Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Total number of urinary incontinence episodes per week

SECONDARY OUTCOMES:
Number of micturition per day, number of urinary urgency episodes per day, volume voided per micturition and QOL

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Development Planning, Study Director — Ono Pharmaceutical Co. Ltd

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401